CLINICAL TRIAL: NCT04745429
Title: Combination of Breathing Exercises, Cold Exposure, and Meditation Mitigate Psoriasis - Open Label, Randomized, Controlled Trial
Brief Title: Non-pharmacological Mitigation of Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jan Czarnecki, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNN/347/18/KE
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis; Stress; Inflammation; Depression; Pruritus; Sleep Disorder; Quality of Life
Keywords: meditation; exposure to cold; inflammation; breathing
MeSH Terms: conditions — Psoriasis; Inflammation; Depression; Pruritus; Sleep Wake Disorders; Respiratory Aspiration | interventions — Breathing Exercises; Meditation

STUDY DESIGN:
Intervention Model Description: Two groups, intervention and control, 10 weeks of intervention. Study visits, blood, saliva collection twice: "before" and "after".
Masking Description: It is impossible to conduct a masked trial as the intervention is collection of exercises that have to be taught by an instructor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 19 people suffering from psoriasis were performing excersises for 10 weeks
  Interventions: Other: breathing exercises, cold exposure and meditation
- Control (No Intervention): 19 people suffeing from psoriasis that didn't train the exercises

INTERVENTIONS:
Other: breathing exercises, cold exposure and meditation — It is a combination of exercises that include breathing exercises, cold exposure and meditation
  Arms: Intervention

SUMMARY:
In the past few years, research has provided evidence for a possibility of dampening immune system by one's will after undergoing a specific training program. Aim of this study was to verity the efficacy in affecting both mind and body by assessing psoriasis activity and psychological functioning. Among the members of both of the groups intensity of skin lesions and pruritus were assessed, consultation regarding treatment took place and multiple questionnaires regarding sleep quality, mindfulness and depressive symptoms were distributed. Blood samples were collected to asses intensity of inflammation, including interleukins.

DETAILED DESCRIPTION:
Psoriasis is a skin disease of an unknown origin. Current understanding of its pathophysiology focuses on an undefined imbalance between the immune system and the nervous system. In this study the researchers assessed the effects of a training program which was proven to affect both. A group of psoriatic patients volunteered, and were randomized to either the intervention (n = 19), or control group (n = 19). Subjects in the intervention group were trained for 10 weeks in breathing techniques, exposure to cold and meditation. The control group was not trained.

After two weeks of the intervention, a full lockdown due to the COVID-19 pandemics was introduced. Modified protocol included exercises possible to conduct at home only.

Two study visits (before and after the intervention) took place.

Total count of variables analysed equaled 60. Primary endpoints regarded intensity of psoriasis. This group included laboratory markers (hsCRP, WBC, LEU, MONO, IL-6, IL-8, IL-10, IL-17, TNFalpha) measured in serum and saliva, visual skin assessment performed by a health professional using Psoriasis Area Severity Index, consultations regarding treatment, and results of the questionnaires (Dermatological Life Quality Index, pruritus). Secondary endpoints pertained comorbidities of psoriasis. These were also assessed using questionnaires, and included Pittsburgh Sleep Quality Index, Patient Health Questionnaire - 9 (depressive symptoms), Five Facet Mindfulness Questionnaire, Perceived Stress Scale - 10.

The intervention is a specific combination of breathing exercises, meditation and cold exposure. It has been previously proven to have an effect among healthy young males who were able to drop febrile temperatures induced with an intravenously distributed LPS. That phenomena was achieved using previously trained breathing techniques.

For 10 weeks members of the intervention group were trained via popular social media platform. Exercises included exposure to cold using regular, cold showers, performing breathing exercises finished with a short meditation session. Length and general difficulty were gradually built up.

Initially, total number of the subjects equaled 54. 31 for the intervention group and 23 for the control group. Due to drop-out or meeting the exclusion criteria, final count for both of the groups was 19 participants.

ELIGIBILITY:
Inclusion Criteria:

* Aforementioned Age
* Confirmed diagnosis of plaque psoriasis

Exclusion Criteria:

* ultraviolet therapy 2 months prior or introduced later during intervention period
* lifestyle changes defined as changing jobs, introducing a new diet, or sport, or changing their place of residence
* kidney disease
* heart disease
* active infection
* pregnancy
* breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index | 10 weeks
  Visual assessment of the skin condition. Extreme values: 0-72. The lower the score, the better
Dermatology Life Quality Index | 10 weeks
  Questionnaire regarding the influence of the disease on everyday functioning. Extreme values: 0-30. The lower the value, the better.
Pruritus Questionnaire | 10 weeks
  Intensity of pruritus measured with a questionnaire. Extreme values 0-18. The lower the score, the better.
Ointment treatment | 10 weeks
  Change in ointment treatment - consultation result
high sensitivity C-reactive protein in serum | 10 weeks
  Levels of C-reactive protein in serum using high sensitivity measurements
Interleukin 6 in serum | 10 weeks
  Level of interleukin 6 in measured serum
Interleukin 6 in saliva | 10 weeks
  Level of interleukin 6 in measured saliva
Interleukin 8 in serum | 10 weeks
  Level of interleukin 8 measured in saliva
Interleukin 8 in saliva | 10 weeks
  Levels of interleukin 8 measured in saliva
Interleukin 10 in serum | 10 weeks
  Levels of interleukin 10 measured in serum
Interleukin 10 in saliva | 10 weeks
  Levels of interleukine 10 measured in saliva
Tumor Necrosis Factor alpha in serum | 10 weeks
  Levels of Tumor Necrosis Factor in serum
Tumor Necrosis Factor alpha in saliva | 10 weeks
  Levels of Tumor Necrosis Factor in saliva
Monocyte count | 10 weeks
  Monocyte count in peripheral blood morphology
Lymphocyte count | 10 weeks
  Lymphocyte count in peripheral blood morphology
Platelet count | 10 weeks
  Platelet count in peripheral blood morphology
Neutrophil count | 10 weeks
  Neutrophil count in peripheral blood morphology

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire - total score | 10 weeks
  Total result of FFMQ. Extreme values: 39 - 195. The higher the score, the better.
Non-Judgement component of the Five Facet Mindfulness Questionnaire | 10 weeks
  Index regarding skill of restraining from labeling. Extreme values: 8-40. The higher the score, the better
Non-Reactivity component of the Five Facet Mindfulness Questionnaire | 10 weeks
  Index measuring skill of restraining from uncontrolled reactions. Extreme values: 7-35. The higher the score, the better
Observation component of the Five Facet Mindfulness Questionnaire | 10 weeks
  Index regarding objective observation. Extreme values: 8-40. The higher the score, the better
Acting with awareness component of the Five Facet Mindfulness Questionnaire | 10 weeks
  Index regarding everyday awareness. Extreme values: 8-40. The higher the score, the better
Describing component of the Five Facet Mindfulness Questionnaire | 10 weeks
  Index regarding skill of objective describing. Extreme values: 8-40. The higher the score, the better
Perceived Stress Scale - 10 | 10 weeks
  Questionnaire regarding everyday stress. Extreme values 0-40. The lower the score, the better.
Patient Health Questionnaire - 9 | 10 weeks
  Questionnaire regarding depressive symptoms. Extreme values 0 - 27. The lower the score, the better
Pittsburgh Sleep Quality Index | 10 weeks
  Questionnaire regarding sleep quality. Extreme values 0 - 21, the lower the score, the better

CONTACTS AND LOCATIONS:
Overall Officials: Anna Zalewska-Janowska, professor, Study Director — Psychodermatology Department
Locations (1):
- Medical Univeristy of Lodz, Chair of Clinical Immunology and Rheumatology, Lodz, Łódź Voivodeship, Poland